CLINICAL TRIAL: NCT02441062
Title: Impact of Ga-68 DOTATOC PET-CT Imaging in Management of Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sue O'Dorisio (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Sue O'Dorisio, Professor, Pediatrics Hematology/Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201503708
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumors; Neuroblastoma; Medulloblastoma
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Neuroblastoma; Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTATOC PET/CT (Other): Study participants will receive 68Ga-DOTATOC and undergo a PET/CT imaging study. Subjects may receive a second 68Ga-DOTATOC PET/CT for restaging after therapy 12-36 months following the first scan.
  Interventions: Drug: 68Ga-DOTATOC PET/CT

INTERVENTIONS:
Drug: 68Ga-DOTATOC PET/CT — Ga-68 DOTATOC PET-CT on management of patients with somatostatin receptor positive tumors

SUMMARY:
Participants in this study have been diagnosed with a tumor such as a carcinoid, neuroendocrine tumor, neuroblastoma, Ewing's sarcoma, or brain tumor that has cells which carry somatostatin receptors.

The purpose of this research study is to see if the tumor can be identified using a special procedure called a positron emission tomography (PET) scan and how the results of this imaging procedure will change the management of the tumor.

DETAILED DESCRIPTION:
This is a prospective, Phase II, single center, open-label study in a total of 200 participants with histologically proven neuroendocrine tumor or other somatostatin receptor positive tumors. Eligible participants will undergo baseline assessments at enrollment. They will receive 68Ga-DOTATOC and undergo a PET/CT imaging study. Participants may receive a second 68Ga-DOTATOC PET/CT for restaging after therapy 12-36 months following the first scan.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 6 months
3. Histologically diagnosed neuroendocrine tumor or other tumor with probable somatostatin receptors subtype 2
4. Karnofsky performance status or Lansky Play Scale status of ≥ 60 (or ECOG/WHO equivalent)
5. Subject is male; or is a female who is either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (> 1 years without menses), ≥60 years old,or of childbearing potential for whom a pregnancy test (with the results known prior to investigational product administration) is negative. A negative pregnancy test will be required for all female subjects with child bearing potential. If a false pregnancy test is suspected, e.g., perimenopausal condition, an obstetrician will be consulted to determine if she is/is not capable of becoming pregnant. Female must also be non-lactating.

Exclusion Criteria:

1. Subject weighs more than 450 pounds. (Subjects who weigh more than 450 pounds will not be able to fit inside the imaging machines) or otherwise cannot be safely fit into the imaging system.
2. Inability to lie still for the entire imaging time (due to cough, severe arthritis, etc.)
3. Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
4. Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance.
5. Peptide receptor radionuclide therapy (PRRT) within 4 weeks of Ga-68 DOTATOC PET/CT scan.
6. Treatment with Sandostatin LAR within 4 weeks, SQ Octreotide within 12 hours, or Lanreotide injection within 8 weeks of Ga-68 DOTATOC PET/CT (+/-5%).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary S O'Dorisio, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menda Y, Ponto LL, Schultz MK, Zamba GK, Watkins GL, Bushnell DL, Madsen MT, Sunderland JJ, Graham MM, O'Dorisio TM, O'Dorisio MS. Repeatability of gallium-68 DOTATOC positron emission tomographic imaging in neuroendocrine tumors. Pancreas. 2013 Aug;42(6):937-43. doi: 10.1097/MPA.0b013e318287ce21. PMID 23587853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 68Ga-DOTATOC PET/CT
Started | 122
Completed | 122
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga-DOTATOC PET/CT
Number analyzed (Participants) | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 98
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 104
  More than one race | 1
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Treatment Management Based on Findings of the Gallium Ga 68-edotreotide PET/CT Scan
Description: Referring physicians will be asked to fill out pre-PET and post-PET scan forms to provide information on the management and treatment strategy of the patient before the PET-CT scan and after the information from the PET-CT study is available. This is the same methodology used in the National Oncologic PET Registry study; change in management strategy criteria are modified for the specific treatment strategies used in NET.
Time Frame: 36 months
Population: Study stopped early, 114 of the 122 patients enrolled were analyzed for outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-DOTATOC PET/CT
Number analyzed (Participants) | 114
Participants
  Major change | 54
  Minor change | 6
  No change | 54

ADVERSE EVENTS:
Time Frame: Adverse events collected at the time of scan, 1 day post scan, and 6-18 months post scan.
Arm/Group | 68Ga-DOTATOC PET/CT
All-Cause Mortality (participants affected / at risk) | 2/122
Serious Adverse Events (participants affected / at risk) | 0/122
Other Adverse Events (participants affected / at risk) | 42/122
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-DOTATOC PET/CT (N=122)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (11)
Vomiting (Gastrointestinal disorders) | 1 (2)
Fever (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 1 (2)
Flushing (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT02441062/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT02441062/Prot_SAP_001.pdf